CLINICAL TRIAL: NCT03943277
Title: Usefulness of White Blood Cell Count (WBCC) During Infection: a Comparison Between Hospitalized Geriatric and Young Groups.
Brief Title: Usefulness of White Blood Cell Count (WBCC) During Infection in Geriatric Patient
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nathalie compté, Clinic head of geriatric unit, Universitair Ziekenhuis Brussel
Other Study IDs: UZCompte1
Record Dates: First submitted 2019-04-25; First posted 2019-05-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: White Blood Cells Engulfing Red Blood Cells
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with infection: Acute inflammation is defined as a CRP ≥ 10 mg/l. We will include 2 groups of participants:
  A group with an inflammatory syndrome and infection; infection being defined as:
  1. Viral infection confirmed by nasopharynx swab for: influenza, RSV, parainfluenza, rhinovirusses, coronavirusses.
  2. Bacterial infection confirmed with positive blood culture, positive articular punction, positive expectorations, pneumonia on chest radiograph, or infection documented by abdominal imagery (CT or echo), a positive urine culture with a confirmed pyelonephritis with a renal echography or a DMSA scintigraphy or specific clinical symptoms for pyelonephritis and positive hemoculture. A positive urine culture alone is not considered as urine infection because of the high prevalence of asymptomatic bacteriuria in geriatric patients.
  Interventions: Other: No intervention, observational study
- patient without infection: Acute inflammation is defined as a CRP ≥ 10 mg/l. We will include 2 groups of participants:
  => B) A group with inflammatory syndrome and inflammatory diseases without infection: defined as:
  1. Confirmed pulmonary embolism (PE) by CT or ventilation-perfusion scintigraphy
  2. Microcrystalline arthritis diagnosed by articular punction
  3. Crush syndrome or rhabdomyolyses defined by history of a fall and raised creatine kinase in blood sample.
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study — No intervention observational study

SUMMARY:
In the general population, increased WBCC and neutrophil count are widely used as markers for infection during inflammatory states 1. However, 32% of geriatric patients with an infection do not develop an increase in WBCC 2. The hypothesis is that with inflammation, geriatric patients have a misadapted response of the immune system (IS) 3.

Our recent retrospective study 4 has shown that total and differential WBCC were not correlated with infection in a geriatric hospitalized population. Therefore, WBCC does not seem to be a reliable marker for infection in geriatric hospitalized patients. The neutrophil/lymphocyte ratio, and CRP, seem to be better markers.

the aim of the study to investigate this hypothesis prospectively and assess the role of aging and chronic diseases (such as cardiovascular diseases (CVD) and risk factors (CVRF) 5, cytomegalovirus (CMV) infection 6, periodontitis 7, onychomycosis 8 ) in this process and assess the role of a geriatric assessment.

To assess the usefulness of WBCC in the diagnosis of infection in geriatric patients and to address the contribution of ongoing chronic co-morbidities and age to WBCC-kinetics during an acute inflammatory syndrome, young and geriatric hospitalized patients with an inflammatory syndrome with and without infection will be compared

DETAILED DESCRIPTION:
Study design Observational prospective study

The subjects Number of subjects 200 subjects: Average value CRP: group 1: 55; group 2: 84 Average standard deviation: 70.52 Power 80%: 158 deelnemers Power 90%: 202 deelnemers alpha = 0.05 2-sample T-test.

Inclusion criteria

Acute inflammation is defined as a CRP ≥ 10 mg/l. We will include 2 groups of participants:

* A) A group with an inflammatory syndrome and infection; infection being defined as:

  1. Viral infection confirmed by nasopharynx swab for: influenza, RSV, parainfluenza, rhinovirusses, coronavirusses.
  2. Bacterial infection confirmed with positive blood culture, positive articular punction, positive expectorations, pneumonia on chest radiograph, or infection documented by abdominal imagery (CT or echo), a positive urine culture with a confirmed pyelonephritis with a renal echography or a DMSA scintigraphy or specific clinical symptoms for pyelonephritis and positive hemoculture. A positive urine culture alone is not considered as urine infection because of the high prevalence of asymptomatic bacteriuria in geriatric patients.
* B) A group with inflammatory syndrome and inflammatory diseases without infection: defined as:

  1. Confirmed pulmonary embolism (PE) by CT or ventilation-perfusion scintigraphy
  2. Microcrystalline arthritis diagnosed by articular punction
  3. Crush syndrome or rhabdomyolyses defined by history of a fall and raised creatine kinase in blood sample.

Exclusion criteria Immunosuppressive therapy (NSAIDs, corticosteroids, chemotherapy, immunotherapy), active cancer, antibiotics before admission, hematological diseases

Replacement of subjects None.

Restrictions and prohibitions for the subjects None.

Procedures

A) Questionnaires:

taken at UZ Brussels

* Social: age, home, sex, marital status.
* Clinical: smoking and alcohol habits, streptococcus pneumoniae and influenza vaccination status, allergies, BMI, medical history, current treatment, reason for current hospitalization.
* Comprehensive geriatric assessment:
* CIRS-G (Cumulative Illness Rating Score): to quantify disease burden. It rates each organ system on a scale of 0 to 4, and differentiates older adults with the highest risk of and severity of infection, from those with lower infection risk. 20
* Katz scale (ADL: assessment of activities of daily living): It rates 6 tasks of daily living (bathing, dressing, toilet, transfer, continence and eating) on a scale from 1 to 4. A low score means absence of dependence, and a high score the maximum of dependence for the task. 21
* MMSE (Mini Mental Status Examination): a 0-30 score of cognitive functions, <24/30 meaning cognitive function impairment. 22 Patients with dementia:the investigators will request approval to be included in the study to the family of the patients.
* MUST (Malnutrition Universal Screening Tool): to assess nutritional status. It divides patients into 3 groups: A low risk of malnutrition (score 0). A medium risk of malnutrition (score 1): then it is recommended to observe the patient for dietary intake. A high risk of malnutrition (score ≥2): treat the malnutrition. 23
* Questionnaire for periodontal health. The newly developed questionnaire produces a reliable assessment of the individual risk of periodontitis (total score) and the need for periodontal treatment as well as the differentiation between gingivits and peridontitis. 24
* Grip strength: Inflammatory states in the elderly are also associated with a decrease in muscle strength and fatigue resistance, as seen at UZ Brussels by Bautmans et al. The reduced strength and fatigue resistance in geriatric patients with inflammation are significantly related with the concentration of circulating CRP levels. 25 In the study, the investigators will use the martin vigorimeter which is at our disposal at the geriatrics ward of UZ Brussels, to measure the patients' grip strength and muscle fatiguability and determine which factors seem to contribute to a decrease in muscle strength (CRP, CVD, CVR, infection, periodontitis, CMV status, onychomycosis, age). the investigators will use the Martin vigorimeter (Elmed, Addison, IL) to assess grip strength and fatiguibility. The investigators will ask the patients to squeeze the rubber bulb of the vigorimeter as hard as possible in 3 consecutive attempts, to assess their grip strength. The highest score for each hand is recorded. Fatigue resistance will be assessed by asking the patient to squeeze the bulb of the vigorimeter as hard as possible and to maintain this pressure as long as possible; the time (seconds) until the pressure diminished to half of the maximal grip strength is recorded for each hand.25 26 B) Collection of data from physical examination C) Clinical evaluation of onychomycosis of the toenails: the investigators will perform a clinical examination of the toenails. Following parameters are found to be significantly related to positive mycology results in onychomycosis patients 8: scaling on one or both soles, white crumbly patches on the nail surface, and an abnormal colour of the nail.

D) Follow up of bacterial and viral culture analyses

Observational data from bacterial and viral samples during hospitatalization :

1. Viral infection confirmed by nasopharynx swab for: influenza, RSV, parainfluenza, rhinovirusses, coronaviruses
2. Bacterial infection confirmed with positive blood culture, positive articular punction, positive expectorations, pneumonia on chest radiograph, or infection documented by abdominal imagery (CT or echo), a positive urine culture with a confirmed pyelonephritis with a renal echography or a DMSA scintigraphy or specific clinical symptoms for pyelonephritis and positive hemoculture. A positive urine culture alone is not considered as urine infection because of the high prevalence of asymptomatic bacteriuria in geriatric patients.

E) Follow up of blood analyses:

Observational data from blood samples during hospitalization:

* Day 0 (at the emergency department): CRP, total and differential WBCC, renal function
* Day 1: at hospitalization, within 24h of admission
* Geriatric patients: CRP, total and differential WBCC, renal function, hepatic function (transaminases), albumin, prealbumin, protein profile and monoclonal protein, vitamin B12, folic acid, hemoglobin, hematocrit, TSH, CMV-serology.
* Young patients: CRP, total and differential WBCC, renal function, albumin, vitamin B12, folic acid, TSH, CMV-serology.
* Day 3: CRP, total and differential WBCC.
* Day 5: CRP, total and differential WBCC.

Flowchart Questionnaires, blood samples: conducted by Hanne Maes. Supervising MD: Dr. Nathalie Compté, UZ Brussels.

Randomisation/blinding Observational study, not applicable.

Prior and concomitant therapy All medication can be continued during this study.

Study analysis Statistical analysis the investigators will perform student t-tests or Mann-Whitney rank sum tests to compare geriatric/young patients with and without infection. To assess the contribution of age, comorbidities and geriatric syndrome in the kinetics of WBCC, the investigators will perform univariate and multivariate analyses.

ELIGIBILITY:
Inclusion Criteria:

Acute inflammation is defined as a CRP ≥ 10 mg/l. We will include 2 groups of participants:

* A) A group with an inflammatory syndrome and infection; infection being defined as:

  1. Viral infection confirmed by nasopharynx swab for: influenza, RSV, parainfluenza, rhinovirusses, coronavirusses.
  2. Bacterial infection confirmed with positive blood culture, positive articular punction, positive expectorations, pneumonia on chest radiograph, or infection documented by abdominal imagery (CT or echo), a positive urine culture with a confirmed pyelonephritis with a renal echography or a DMSA scintigraphy or specific clinical symptoms for pyelonephritis and positive hemoculture. A positive urine culture alone is not considered as urine infection because of the high prevalence of asymptomatic bacteriuria in geriatric patients.
* B) A group with inflammatory syndrome and inflammatory diseases without infection: defined as:

  1. Confirmed pulmonary embolism (PE) by CT or ventilation-perfusion scintigraphy
  2. Microcrystalline arthritis diagnosed by articular punction
  3. Crush syndrome or rhabdomyolyses defined by history of a fall and raised creatine kinase in blood sample.

Exclusion Criteria:

Immunosuppressive therapy (NSAIDs, corticosteroids, chemotherapy, immunotherapy), active cancer, antibiotics before admission, hematological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Young and older patient with an inflammatory syndrome (CRP > 10 mg/dl) with or without infection
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Usefulness of white blood cell count (WBCC) during infection in geriatric patient | 1.5 years
  observation of WBCC is correlated with infection by older patient
Delta of wbcc | 1.5 years
  the significance of a Delta of WBCC (Delta= □((White blood cell count during acute infection or acute inflammatory events)/(White blood cell count in chronic circumstances)) ) in geriatric patients with acute infections or inflammatory events

CONTACTS AND LOCATIONS:
Overall Officials: Compté Nathalie, Dr, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
data will be maybe described in an article

REFERENCES:
- [Result] Compte N, Dumont L, Bron D, De Breucker S, Praet JP, Bautmans I, Pepersack T. White blood cell counts in a geriatric hospitalized population: A poor diagnostic marker of infection. Exp Gerontol. 2018 Dec;114:87-92. doi: 10.1016/j.exger.2018.11.002. Epub 2018 Nov 6. PMID 30412726
- [Result] Compte N, Bailly B, De Breucker S, Goriely S, Pepersack T. Study of the association of total and differential white blood cell counts with geriatric conditions, cardio-vascular diseases, seric IL-6 levels and telomere length. Exp Gerontol. 2015 Jan;61:105-12. doi: 10.1016/j.exger.2014.11.016. Epub 2014 Nov 22. PMID 25446500

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03943277/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03943277/ICF_001.pdf